CLINICAL TRIAL: NCT02740933
Title: Demeclocycline Fluorescence for Intraoperative Delineation Brain Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, William T. Curry, MD, William T. Curry, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-280
Record Dates: First submitted 2016-03-15; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Brain Tumor
Keywords: Brain Tumor Surgery
MeSH Terms: conditions — Brain Neoplasms | interventions — Demeclocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Demeclocycline (Experimental): All subjects will take Demeclocycline 300 mg po bid. Patients will be advised to take demeclocycline on an empty stomach, at least 1-2 hours before meals, and they will be warned that it can reduce the efficacy of oral contraceptives.
  The investigators will begin by treating subjects with 2 days of demeclocycline. The investigators will increase the numbers of days that subjects are exposed to demeclocycline in increments of 1 day until at least 80% of patients at a given dose have detectably fluorescent tumors, or participants reach 5 days of drug, whichever comes first.
  Interventions: Drug: Demeclocycline

INTERVENTIONS:
Drug: Demeclocycline
  Other Names: Declomycin

SUMMARY:
This research study is studying a drug called Demeclocycline that may help brain surgeons see tumors with a microscope during surgery.

DETAILED DESCRIPTION:
This research study is a Feasibility Study, which is the first time investigators are examining this study intervention.The FDA (the U.S. Food and Drug Administration) has not approved Demeclocycline for your specific disease but it has been approved for other uses.

In this research study, the investigators would like to determine the lowest dose of Demeclocycline that will allow surgeons to detect tumor cells during surgery. These cells will be marked through a process called fluorescence, which will cause tumor cells to glow brightly on an image in comparison to its surroundings.

ELIGIBILITY:
Inclusion Criteria:

* Participants must present with a gadolinium-enhancing brain lesion (or lesions) that are thought by the neuroradiologist and the neurosurgeon to be consistent with high-grade glioma. These may be newly diagnosed lesions or recurrent tumors.
* The patient must not be pregnant or nursing. Tetracycline (Demeclocycline, Doxycycline, Minocycline, Tetracycline, and Tigecycline) are classified as FDA pregnancy category D. Maternal ingestion of Tetracyclines during pregnancy may cause tooth discoloration, enamel defects, and other congenital anomalies. Tetracyclines are excreted in human breast milk; however, the extent of absorption of Tetracyclines by the breastfed infant is not known.
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥ 3,000/mcL
  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤ 4 × institutional upper limit of normal
  * creatinine < 2mg/dL
* Ability to understand and the willingness to sign a written informed consent document.
* Participants must be undergoing a surgical procedure with the intention of removing more tissue than what would be taken for a biopsy.

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Demeclocycline.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or nursing women are excluded from this study because Demeclocycline is a known Teratogenic agent, pregnancy category D. It is known to be excreted in breast milk.
* Patients taking etinoid medications by mouth (such as Acitretin, Isotretinoin), Strontium Ranelate may not take Demeclocycline because of toxic interactions
* Patients taking any tetracycline class of drug (i.e. Minocycline, etc).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Detectable fluorescence in brain tumors by confocal microscopy after oral dosing of demeclocycline (Y/N). | 2 years
  Detectable fluorescence via confocal microscopy

SECONDARY OUTCOMES:
Sensitivity And Specificity Of Demeclocycline-Enhanced Multimodal Confocal Microscopy of Excised Glioma Specimens | 2 years
  We aim to measure the sensitivity and specificity with which tumors can be diagnosed accurately after satisfactory detection of fluorescence

CONTACTS AND LOCATIONS:
Overall Officials: William T Curry, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to present on and publish the data acquired from this study.

REFERENCES:
- [Background] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895
- [Background] Pichlmeier U, Bink A, Schackert G, Stummer W; ALA Glioma Study Group. Resection and survival in glioblastoma multiforme: an RTOG recursive partitioning analysis of ALA study patients. Neuro Oncol. 2008 Dec;10(6):1025-34. doi: 10.1215/15228517-2008-052. Epub 2008 Jul 30. PMID 18667747
- [Background] Sanai N, Polley MY, McDermott MW, Parsa AT, Berger MS. An extent of resection threshold for newly diagnosed glioblastomas. J Neurosurg. 2011 Jul;115(1):3-8. doi: 10.3171/2011.2.jns10998. Epub 2011 Mar 18. PMID 21417701
- [Background] McGirt MJ, Mukherjee D, Chaichana KL, Than KD, Weingart JD, Quinones-Hinojosa A. Association of surgically acquired motor and language deficits on overall survival after resection of glioblastoma multiforme. Neurosurgery. 2009 Sep;65(3):463-9; discussion 469-70. doi: 10.1227/01.NEU.0000349763.42238.E9. PMID 19687690
- [Background] Laws ER, Parney IF, Huang W, Anderson F, Morris AM, Asher A, Lillehei KO, Bernstein M, Brem H, Sloan A, Berger MS, Chang S; Glioma Outcomes Investigators. Survival following surgery and prognostic factors for recently diagnosed malignant glioma: data from the Glioma Outcomes Project. J Neurosurg. 2003 Sep;99(3):467-73. doi: 10.3171/jns.2003.99.3.0467. PMID 12959431
- [Background] Stummer W, Reulen HJ, Meinel T, Pichlmeier U, Schumacher W, Tonn JC, Rohde V, Oppel F, Turowski B, Woiciechowsky C, Franz K, Pietsch T; ALA-Glioma Study Group. Extent of resection and survival in glioblastoma multiforme: identification of and adjustment for bias. Neurosurgery. 2008 Mar;62(3):564-76; discussion 564-76. doi: 10.1227/01.neu.0000317304.31579.17. PMID 18425006
- [Background] Liu JT, Meza D, Sanai N. Trends in fluorescence image-guided surgery for gliomas. Neurosurgery. 2014 Jul;75(1):61-71. doi: 10.1227/NEU.0000000000000344. PMID 24618801
- [Background] Senft C, Bink A, Franz K, Vatter H, Gasser T, Seifert V. Intraoperative MRI guidance and extent of resection in glioma surgery: a randomised, controlled trial. Lancet Oncol. 2011 Oct;12(11):997-1003. doi: 10.1016/S1470-2045(11)70196-6. Epub 2011 Aug 23. PMID 21868284
- [Background] Zehri AH, Ramey W, Georges JF, Mooney MA, Martirosyan NL, Preul MC, Nakaji P. Neurosurgical confocal endomicroscopy: A review of contrast agents, confocal systems, and future imaging modalities. Surg Neurol Int. 2014 Apr 28;5:60. doi: 10.4103/2152-7806.131638. eCollection 2014. PMID 24872922
- [Background] Sanai N, Snyder LA, Honea NJ, Coons SW, Eschbacher JM, Smith KA, Spetzler RF. Intraoperative confocal microscopy in the visualization of 5-aminolevulinic acid fluorescence in low-grade gliomas. J Neurosurg. 2011 Oct;115(4):740-8. doi: 10.3171/2011.6.JNS11252. Epub 2011 Jul 15. PMID 21761971
- [Background] Wirth D, Snuderl M, Sheth S, Kwon CS, Frosch MP, Curry W, Yaroslavsky AN. Identifying brain neoplasms using dye-enhanced multimodal confocal imaging. J Biomed Opt. 2012 Feb;17(2):026012. doi: 10.1117/1.JBO.17.2.026012. PMID 22463044
- [Background] Snuderl M, Wirth D, Sheth SA, Bourne SK, Kwon CS, Ancukiewicz M, Curry WT, Frosch MP, Yaroslavsky AN. Dye-enhanced multimodal confocal imaging as a novel approach to intraoperative diagnosis of brain tumors. Brain Pathol. 2013 Jan;23(1):73-81. doi: 10.1111/j.1750-3639.2012.00626.x. Epub 2012 Aug 28. PMID 22882328
- [Background] Wirth D, Snuderl M, Curry W, Yaroslavsky A. Comparative evaluation of methylene blue and demeclocycline for enhancing optical contrast of gliomas in optical images. J Biomed Opt. 2014 Sep;19(9):90504. doi: 10.1117/1.JBO.19.9.090504. PMID 25239672